CLINICAL TRIAL: NCT01821001
Title: Vaginal Bromocriptine for the Treatment of Adenomyosis
Brief Title: Vaginal Bromocriptine for Treatment of Adenomyosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elizabeth A. Stewart, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-007353
Record Dates: First submitted 2013-03-21; First posted 2013-03-29 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Adenomyosis
Keywords: Adenomyosis; Dysmenorrhea; Abnormal Uterine bleeding; Heavy Menstrual Bleeding; Menorrhagia
MeSH Terms: conditions — Adenomyosis; Dysmenorrhea; Metrorrhagia; Menorrhagia | interventions — Bromocriptine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaginal Bromocriptine (Experimental): Patients will receive 2.5 mg of vaginal bromocriptine tablet twice a day for the intervention. This will be administered for 6 months.
  Interventions: Drug: Vaginal Bromocriptine

INTERVENTIONS:
Drug: Vaginal Bromocriptine — Patients will receive 2.5 mg of vaginal bromocriptine tablet twice a day for the intervention. This will be administered for 6 months.
  Other Names: Cycloset; Parlodel

SUMMARY:
Adenomyosis is a rare non-malignant disease of the uterus that causes significant symptoms including heavy menstrual bleeding and pelvic pain. The only widely accepted treatment for adenomyosis is hysterectomy. The investigators will use a dopamine agonist, bromocriptine, as a therapy based on animal models of the disease and our prior clinical research to observe any objective improvement in the extent of the disease using Magnetic Resonance Imaging (MRI)and standard measurements for other gynecologic diseases to measure symptomatology.

DETAILED DESCRIPTION:
Women with adenomyosis proven with MRI will be considered for the intervention with bromocriptine. They will be reassessed at 1, 6 and 9 months. Patients will get a stipend for each visit they complete. The study will end for the enrolled subject at 9th month follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Women able to give informed consent and willing and able to attend all study visits
2. Premenopausal women at least 25 years of age
3. No evidence of High Grade SIL by pap smears or HPV testing within institutional guidelines
4. MRI or ultrasound imaging consistent or highly suggestive of adenomyosis
5. Use of barrier contraception, sterilization or sexual abstinence

Exclusion Criteria:

1. Women actively trying for pregnancy, currently pregnant, less than six months postpartum or breastfeeding
2. Uterine size > 20 weeks
3. Active pelvic infection or current use of intrauterine contraceptive device
4. Current use of GnRH agonists or antagonists, or contraceptive steroids
5. MRI suggestive of malignant disease of uterus, ovary, or cervix
6. Hypersensitivity to bromocriptine or ergot alkaloids
7. History of gastrointestinal ulcers
8. History of syncope, syncopal migraine or seizure
9. Uncontrolled hypertension
10. History of myocardial infarction, uncontrolled hypertension, heart valve disorder or cerebrovascular accident
11. History of diabetes mellitus except gestational diabetes
12. History of Parkinson's Disease
13. History of psychosis
14. History of pleural or pericardial effusion
15. History of pulmonary fibrosis or thickening of the pleura
16. History of lactose intolerance
17. History of Reynaud's Disease
18. Use of opioid pain medications

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Objective improvement of adenomyosis | 6 months
  All patients will get a baseline imaging of the uterus with MRI and a brief procedure, similar to a pap smear, to obtain tissue from the uterus and also a blood draw. Patients will then receive vaginal bromocriptine twice daily and will be reassessed at 6 months with an MRI to see objective improvement in the extent of the disease. This 6 month visit is the only one that would require an in person visit to the research site (Mayo Clinic in this case)

SECONDARY OUTCOMES:
Scores from questionnaires that assess the severity of symptoms from adenomyosis | 9 months
  Patients will fill out questionnaires at 1, 3, 6 and 9 months. These questionnaires are validated for study of gynecologic diseases and assess the severity of symptoms in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stewart, MD, Principal Investigator — Mayo Clinic; Zaraq Khan, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States